CLINICAL TRIAL: NCT05107791
Title: Effects of Stulln Eye Drops and Accommodative Training on Accommodative Responses and Visual Fatigue
Brief Title: Effects of Stulln and Accommodative Training
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: unable to attend the drug for study
Sponsor: Pacific University (Other)
Responsible Party: Principal Investigator, Shun-nan Yang, Director of Vision Performance Institute, Pacific University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Stulln-1
Record Dates: First submitted 2018-02-28; First posted 2021-11-04 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Accommodation Disorder; Visual Fatigue
MeSH Terms: conditions — Asthenopia | interventions — Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stulln Eyedrops (Experimental): Augentropfen Stulln Mono Eye Drops (Stulln eyedrops) will be provided to participants in individual single-use vials. Participants will apply the drops to the two eyes 3 times a day, six days a week before sustained eye use (except Sunday).
  Interventions: Drug: Stulln Eyedrops
- Theta Tears (Sham Comparator): Thera Tears (Sodium Carboxymethylcellulose 0.25%) will be provided to participants in individual single-use vials. Participants will apply the drops to the two eyes 3 times a day, six days a week before sustained eye use (except Sunday).
  Interventions: Drug: Thera Tears

INTERVENTIONS:
Drug: Stulln Eyedrops — Stulln eyedrops will be applied to the anterior surface of cornea 3 times a day, 6 days a week. Half of participants (46) also receive accommodative training during the second stage (month) of the study while the rest maintains the Stulln eyedrops intervention.
  Other Names: Accommodative training
  Arms: Stulln Eyedrops
Drug: Thera Tears — The eyedrops will be used in the identical manner as Stulln eyedrops.
  Arms: Theta Tears

SUMMARY:
The present study tests the hypothesis that Stulln eyedrops improve accommodative functions by improving the short term facility of ciliary muscles that can be transferred into long-term adaptation. To test this, the investigators propose to conduct a prospective randomized control trials where participants with accommodative dysfunctions are randomly assigned to four groups: control, Stulln only and Stulln plus vision training. The investigators' theory predicts that the efficacy of Stulln will be augmented by vision training.

DETAILED DESCRIPTION:
Accommodation is the process of adjusting focal distance to achieve a clear retinal vision by altering the shape of human crystalline lens in the eye. Accommodative responses are composed of two parts, phasic and tonic. The adequate phasic accommodation is needed to form a clear retinal image of near stimuli. The proper tonic accommodation is needed to maintain clear retinal vision after the initial phasic response. The phasic and tonic accommodative responses are mediated by the sympathetic and parasympathetic systems. Accommodative accuracy and endurance is achieved by modifying the neuromuscular connection through repetitive learning and adaptation.

Vision training has been shown effective to increase accommodative amplitude and endurance. Its efficacy is achieved by gradually increasing the difficulty of tasks that require patients to attentively process visual cues to adapt their accommodative responses. Its end goal is to induce effective and permanent adaptations to the visual environment. The process of vision training has been theorized as a bioengineering model in which the neuromuscular signal is altered through visuomotor feedback. The increase in accommodative accuracy is thought to reflect the gain of accommodative responses and the increase of accommodative endurance is the result of maintained tonic neural output.

Empirical studies have shown the Digitalisglycosides (DGS) can enhance muscular contraction and Esculin improves micro vascular circulation. Stulln eyedrops include these active ingredients and have been approved to treat visual discomfort and retinal macular diseases in Europe and China. It also has a very good safety record, without any report of adverse effects to human body for the millions of users each year. The efficacy of Stulln in treating visual discomfort might have resulted from the improved microcirculation of blood and wastes, leading to better ciliary functions. Indeed, empirical studies have shown Stulln application can improve accommodative amplitude, facility and endurance. However, Stullen itself might not produce long-term changes in neuromuscular innervation, as its ingredients can be removed from the human body within an day.

The present study tests the hypothesis that Stulln eyedrops improve accommodative functions by improving the short term accommodative facility and endurance. To test this, the investigators propose to conduct a prospective randomized control trials where participants with accommodative dysfunctions are randomly assigned to three groups: control, Stulln only and Stulln plus vision training. The investigators' theory predicts that the efficacy of Stulln will be augmented by vision training.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 45 years of age.
* Have normal/corrected-to-normal monocular acuity of better than 20/25 for both eyes.
* Have normal contrast sensitivity.
* Be a native English speakers or possess college-level English reading proficiency.
* Have a current optical prescription (obtained less than 2 years ago).
* Have accommodative dysfunctions, including reduced accommodative amplitude, range, facility and endurance.

Exclusion Criteria:

* Have no prismatic correction.
* No clinically significant ocular pathology (e.g., cataract, keratoconus, dry eye, diabetic retinopathy, or age-related macular degeneration) that would limit the effectiveness of vision training.
* Have no binocular dysfunction, including amblyopia, strabismus, and other binocular diseases that would impede accommodative training.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Accommodative amplitude | Baseline, 4th and 8th week
  The change in the diopter value of the closest distance at which the visual image con be kept clear between the baseline, 4-week, and 8-week assessments.
Chang in Accommodative Facility | Baseline, 4th and 8th week
  Change in the frequency of clearing the image with +/- 2D flipper in a minute between the baseline, 4-week, and 8-week assessments.
Change in Accommodative Endurance | Baseline, 4th, and 8th week
  The change in the difference in the frequency of clearing the image in two consecutive minutes measured at the baseline, 4th week, and 8th week.
Change in Visual Fatigue | Baseline, 4th, and 8th week
  Change in the score measured from CISS questionnaire between the baseline, 4-week, and 8-week assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Vision Performance Institute, Forest Grove, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.